CLINICAL TRIAL: NCT06950008
Title: Feasibility Testing of a Patient Navigation Intervention to Improve Risk Management Among Women at High Risk of Breast Cancer
Brief Title: A Patient Navigation Intervention for the Improvement of Risk Management Among Women at High Risk of Breast Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Tasleem Juana Padamsee, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: OSU-24198; NCI-2025-01592 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); R21CA271070 (NIH)
Record Dates: First submitted 2025-03-26; First posted 2025-04-29 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms | interventions — Early Intervention, Educational; Educational Status; Methods; Patient Navigation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (informational websites, PN) (Experimental): Participants receive links to informational websites on breast cancer risk and risk management options on study. Participants also receive phone calls from a single patient navigator and discuss breast cancer risk and risk-management options once a month for 8 months. Participants may choose to receive additional patient navigator phone calls as needed on study.
  Interventions: Other: Educational Intervention; Behavioral: Patient Navigation; Other: Survey Administration; Behavioral: Telephone-Based Intervention
- Arm II (informational websites) (Active Comparator): Participants receive links to informational websites on breast cancer risk and risk management options on study.
  Interventions: Other: Educational Intervention; Other: Survey Administration

INTERVENTIONS:
Other: Educational Intervention — Receive links to informational websites
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
Behavioral: Patient Navigation — Receive patient navigator phone calls
  Other Names: Patient Navigator Program
  Arms: Arm I (informational websites, PN)
Other: Survey Administration — Ancillary studies
Behavioral: Telephone-Based Intervention — Receive patient navigator phone calls
  Arms: Arm I (informational websites, PN)

SUMMARY:
This clinical trial studies whether a patient navigation (PN) intervention can be used to improve risk management among women at high risk of breast cancer. Women with a family history of breast cancer have a higher lifetime risk of developing it. Risk management can benefit women at high risk of breast cancer and can include surveillance routines, preventative surgeries, and medications that can dramatically lower the risk of breast cancer and allow early detection. Although risk management can benefit women at high risk of breast cancer, only a small amount actually use it. PN is a healthcare service that is designed to guide a patient through the healthcare system and reduce barriers to timely screening, follow-up, diagnosis, treatment, and supportive care. The PN intervention in this study is designed to help give women the information and support they need to make choices about their breast cancer risk that they feel good about, which may improve risk management.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Test the feasibility of the PN intervention and of recruiting participants to a randomized controlled trial of the intervention.

OUTLINE: Participants are randomized to 1 of 2 arms.

ARM I: Participants receive links to informational websites on breast cancer risk and risk management options on study. Participants also receive phone calls from a single patient navigator and discuss breast cancer risk and risk-management options once a month for 8 months. Participants may choose to receive additional patient navigator phone calls as needed on study.

ARM II: Participants receive links to informational websites on breast cancer risk and risk management options on study.

After completion of study intervention, participants are followed for up to 1 month.

ELIGIBILITY:
Inclusion Criteria:

* Are non-Hispanic Black or non-Hispanic white
* Identify as women
* Are between 18 and 75 years old
* Have been identified as at potentially high risk by a population-based risk screening program
* Have never been diagnosed with breast or ovarian cancer
* Are early in their risk-management adoption process, defined as currently identifying with stage 0 (never heard of it) or 1 (haven't decided) of the risk-management adoption pathway (R-MAP) in relation to at least one of the four risk-management actions recommended for all high-risk women: attending genetic counseling appointment, having a personalized risk assessment, undergoing annual clinical breast exams, and considering chemoprevention
* Who do not believe cancer can be prevented and/or have not received risk-management guidance from a specialist

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2026-01-10 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Participant satisfaction with patient navigation (PN) intervention (Feasibility) | Up to 9 months
  Will be measured using previously validated survey questions related to patient navigation interactions. Will be defined as at least 50% of intervention arm participants are "satisfied" or "very satisfied" with the PN intervention. Will be formally assessed using a point estimate and 95% one-sided (score-based) confidence interval.
Demand measures (Feasibility) | Up to 9 months
  Measures the use of the patient navigator (PN). Will check that at least 50% of the sample interacted with the patient navigator for a total of at least 15 minutes.
Implementation of PN intervention (Feasibility) | Up to 9 months
  Number of calls and patient navigator (PN contacts.
Practicality of PN intervention (Feasibility) | Up to 9 months
  Percentage of participants that assess the intervention as appropriate and are willing to recommend it for similar others.
Percentage of recruited individuals who eventually enroll (Feasibility) | Up to 6 months
  Will be tracked to help determine the feasibility of attracting appropriate sample sizes to power a later effectiveness-oriented randomized controlled trial. Recruitment success will be indicated by enrollment of ≥ 20% recruited patients and a total of 75 in 6 months. Point estimates for other key measures will be used as supporting evidence of intervention feasibility.
Risk-management adoption pathway (R-MAP) progress | Baseline up to 9 months
  Will descriptively estimate progress in R-MAP stage for each recommended risk-management action, as well as estimate change in other R-MAP measures between baseline and final surveys. Differences in R-MAP progress and other measures described will be estimated between arms at the final time point. Will regard the intervention as worthy of further effectiveness testing if the difference in R-MAP stage between intervention and control arm participants is ≥ .5 points (on the 6-point measurement scale) and ≥ 15% for at least one risk-management action.
Perceived Breast Cancer Risk | Up to 9 months
  The percentage of participants with perceived breast cancer risk indicated by survey responses will be summarized.
Cancer Worry | Up to 9 months
  The percentage of participants with cancer worry indicated by survey responses will be summarized.
Confidence in Coping with Breast Cancer Risk | Up to 9 months
  The percentage of participants with confidence in coping with breast cancer risk indicated by survey responses will be summarized.
Belief that Breast Cancer Risk can be Reduced | Up to 9 months
  The percentage of participants with belief that their breast cancer risk can be reduced indicated by survey responses will be summarized.
Mental Health | Up to 9 months
  Will be assessed via a 5-item inventory at baseline and final surveys.
Information usage (Self-reported) | Up to 9 months
  Self-reported usage of the provided informational websites by the control group will be measured. Number of visits to the informational websites will be summarized.
Information usage (Machine-recorded) | Up to 9 months
  Machine-recorded usage of the provided informational websites by the control group will be measured. Usage will be recorded by tracking the use of the bitly links provided. The number of visits to each informational website will be summarized.

CONTACTS AND LOCATIONS:
Overall Officials: Tasleem J Padamsee, PhD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu